CLINICAL TRIAL: NCT01805869
Title: Oral Specimen and Data Acquisition Study of Subjects Requiring Third Molar Removal
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130033; 13-D-0033
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-07-30

CONDITIONS: Stomatognatic; Tooth Diseases; Diseases; Tooth; Tooth Impaction
Keywords: Third Molar; Specimen Acquisition; Natural History
MeSH Terms: conditions — Tooth Diseases; Disease; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Male or female ages 16-50

SUMMARY:
Background:

- The third molars (wisdom teeth) normally grow in during late adolescence or early adulthood. Many people need or choose to have these teeth removed with oral surgery. Normally, the removed teeth and tissue are thrown away as medical waste. However, oral health researchers want to collect the teeth and tissue for research. They also want to encourage dentists at the National Institutes of Health to improve their skills in oral surgery. This study will collect the teeth and tissue of people who need to have oral surgery to remove their wisdom teeth.

Objectives:

* To provide continued dental skills training for dentists at the National Institutes of Health.
* To collect teeth and tissue samples following wisdom tooth removal surgery.

Eligibility:

- Individuals between 16 and 50 who need to have their wisdom teeth removed.

Design:

* This study will involve a minimum of three visits. There will be a screening visit, a surgery visit, and at least one follow-up visit.
* Participants will be screened with a physical exam and medical history. A full dental exam with x-rays will be given to evaluate the need for surgery.
* At the second visit, participants will have oral surgery to remove their wisdom teeth. The teeth and tissue removed during the surgery will be collected for study.
* Participants will receive drugs to control the pain after surgery. They will also be able to contact a dentist if there are any problems.
* Between 7 and 21 days after surgery, participants will have a followup visit to check the healing. If they are having no problems, this will be the last visit. If there are any postsurgery issues, they will be scheduled for additional visits as needed.

DETAILED DESCRIPTION:
Objective

The objective of this protocol is to collect data and surgical waste tissue for research purpose in subjects undergoing clinically indicated wisdom teeth extraction at the NIH NIDCR Dental clinic with the aim of obtaining generalizable knowledge about oral health while utilizing surgical waste tissue for research studies.

Study Population

The protocol will enroll a convenience sample of 10,000 subjects ages greater than or equal to 16-50 in need of clinically indicated extraction of third molars.

Design

This is a data collection and specimen acquisition protocol. Data and oral tissue samples will be collected for research purpose in subjects undergoing extraction of third molar teeth at the NIH NIDCR dental clinic. If trends in data emerge that warrant further exploration, outcome measures will be identified, and IRB approval or determination of exemption will be requested to carry out the project. Oral specimens removed during a third molar extraction will be distributed for research with appropriate IRB approval.

Subjects will report to the NIH NIDCR dental clinic for 3 visits. The first visit will be a screening evaluation to determine protocol eligibility. Eligible subjects will return for a second visit for the third molar extraction procedure. The third visit will be scheduled approximately 3-40 days after surgery for a post-operative clinical evaluation. Additional visits for standard of care follow up or treatment may be required based on clinical status of subject after surgery.

Outcome Measures

Data collection includes demographics, medical/dental history, examination findings, pain management, medication regimen, adverse events and other data collected from all standard of care procedures.

Oral specimens removed during third molar extraction may include teeth, alveolar bone, excessive gingival tissue and other waste tissue and will be distributed for research as directed by IRB and OHSRP approval for sharing.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages greater than or equal to 16-50 years
* Clinical evidence of need for third molar extraction as determined by medical, dental, and radiographic evaluation by a NIDCR oral surgeon
* Willing to allow for the collection of extracted waste tissue (e.g., teeth, alveolar bone, excessive gingival tissue) to be used for research
* In good general health as defined by the American Society of Anesthesiologists (ASA) status I or II
* Able to understand and sign an informed consent

EXCLUSION CRITERIA:

* Pregnant or nursing women
* Unable to have third molar extraction as determined by NIDCR surgeon/dentist, due to medical conditions (beyond ASA I or II), complexity of the surgery, or history that precludes safe outpatient conscious sedation. These clinical decisions will be based on the risks and benefits related to the surgery.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The protocol will enroll a convenience sample of 10,000 subjects ages >16-50 in need of clinically indicated extraction of third molars.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-06-19 (Actual); Primary Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
data collection | 16 years
  If trends emerge that warrant further exploration, outcome measures will be described

CONTACTS AND LOCATIONS:
Overall Officials: Janice S Lee, DDS, MD, Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-D-0033.html